CLINICAL TRIAL: NCT06151093
Title: Investigating the Effects of Video-Based Balance Games and Balance Exercises on Visual-Spatial Attention With EEG Brain Oscillations
Brief Title: The Effect of Balance Exercises on Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, yasin yildirim, Physiotherapist, MSc, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: E-10840098-772.02.7781
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: EEG Brain Oscillations; Balance Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-based balance games group (Experimental)
  Interventions: Other: Video-based games intervention
- Balance exercises group (Experimental)
  Interventions: Other: Balance exercises

INTERVENTIONS:
Other: Video-based games intervention — These games are applied via using Nintendo Wii
  1st - 2nd Week Applications
  * Basic Step
  * Penguin slide (right-left weight transfer)
  * Snowball flight (right-left weight transfer)
  * Tilt city (right-left weight transfer)
    3rd-4th Week Applications
  * Advanced Step
  * Snowball flight (right-left weight transfer)
  * Penguin slide (right-left weight transfer)
  * Table tilt (weight transfer in 4 directions)
    5th-6th Week Applications
  * Advanced Step
  * Table tilt (weight transfer in 4 directions)
  * Balance bubble (weight transfer to 4 directions)
  * Ski slalom (weight transfer in 4 directions)
  Arms: Video-based balance games group
Other: Balance exercises — 1st-2nd Week Applications On a flat-hard surface;
  * Standing on 2 legs
  * Stepping forward and backward (separately for both feet)
  * Getting into the tandem position and maintaining the position (separately for both feet)
  * Standing on one leg (separately for both feet)
  * Weight transfer in four directions
  * Taking a step back towards the step
  * Stepping on the stability ball
    3rd-4th Week Applications All exercises which applied in 1st and 2nd week are applied on mat.
    5th-6th Week Applications On the balance board;
  * Standing on 2 legs
  * Stepping forward and backward (separately for both feet)
  * Getting into the tandem position and maintaining the position (separately for both feet)
  * Standing on one leg (separately for both feet)
  * Weight transfer in four directions
  * Catching balls thrown by the enforcer
  Arms: Balance exercises group

SUMMARY:
The aim of our study is to examine the effects of balance exercises performed in virtual and real environments on visual-spatial attention and mental rotation in healthy young adult individuals using EEG brain oscillations.

ELIGIBILITY:
Inclusion Criteria:

* There wouldn't be any neurological conditions
* There wouldn't be drug use such as psychiatric drug
* There wouldn't be lower extremity surgery
* There wouldn't be epilepsy
* Be healthy
* Take minimum 68 points of System Usability Scale

Exclusion Criteria:

* Neurologic disorder
* Epilepsy
* Active sport life
* Colour blindness

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
EEG - event related oscillations | Baseline-6 week
  In our research, EEG recordings will be made with the Brain Vision Recorder (Brainproduct, Munich, Germany) device. Recording will be made on 30 channels with 0.1-250 Hz band pass and 500 sample rate features. An elastic cap with 32 Ag-AgCl electrode placement will be used as the cap. The placement of electrodes will be made according to the international 10-20 system and includes FP1, FP2, F7, F3, FZ, F4, F8, FT7, FC3, FCZ, FC4, FT8, T7, C3, CZ, C4, T8, TP7, CP3, CPZ. Recordings will be taken from the electrodes CP4, TP8, P7, P3, PZ, P4, P8, O1, OZ and O2. Additionally, two connected electrodes (A1+A2) will be placed on the front of both earlobes as a reference, and the ground electrode will be placed on the back of the right earlobe. In addition, electrodes placed in the medial upper part and lateral orbital part of the left eye will be used for EOG recording. During shooting, care will be taken to ensure that the impedance values of the electrodes are below 10 kΩ.

CONTACTS AND LOCATIONS:
Overall Officials: Bahar Güntekin, Prof. Dr., Study Director — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No